CLINICAL TRIAL: NCT00953706
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate the Safety and Efficacy of VX-770 in Subjects Aged 12 Years and Older With Cystic Fibrosis Who Are Homozygous for the F508del-CFTR Mutation
Brief Title: Study of Ivacaftor in Cystic Fibrosis Subjects Aged 12 Years and Older Homozygous for the F508del-CFTR Mutation
Acronym: DISCOVER
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Following review of results obtained from a pre-specified 6-month analysis of Part B data the study was terminated on the basis of futility.
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VX08-770-104; 2009-010261-23 (EudraCT Number)
Record Dates: First submitted 2009-08-04; First posted 2009-08-06 (Estimated); Results first posted 2012-08-21 (Estimated); Last update posted 2015-09-11 (Estimated); Status verified 2015-08

CONDITIONS: Cystic Fibrosis
Keywords: Fibrosis; Pancreatic Diseases; Digestive System Diseases; Lung Diseases; Respiratory Tract Diseases; Genetic Diseases, Inborn; Infant, Newborn, Diseases; Pathologic Processes
MeSH Terms: conditions — Cystic Fibrosis; Fibrosis; Pancreatic Diseases; Digestive System Diseases; Lung Diseases; Respiratory Tract Diseases; Genetic Diseases, Inborn; Infant, Newborn, Diseases; Pathologic Processes | interventions — ivacaftor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo matched to ivacaftor tablet orally every 12 hours (q12h) for 16 weeks during Part A (double-blind treatment period), followed by ivacaftor 150 mg tablet orally q12h for 96 weeks during Part B (open-label extension period).
  Interventions: Drug: Ivacaftor; Drug: Placebo
- Ivacaftor (Experimental): Ivacaftor 150 milligram (mg) tablet orally q12h for 16 weeks during Part A (double-blind treatment period), followed by ivacaftor 150 mg tablet orally q12h for 96 weeks during Part B (open-label extension period).
  Interventions: Drug: Ivacaftor

INTERVENTIONS:
Drug: Ivacaftor — Tablet
  Other Names: VX-770
Drug: Placebo — Tablet
  Arms: Placebo

SUMMARY:
The purpose of this study was to evaluate the safety and efficacy of ivacaftor in participants with cystic fibrosis (CF) who were aged 12 years or older and were homozygous for the F508del-CF transmembrane conductance regulator (CFTR) mutation. Ivacaftor is a potent and selective CFTR potentiator of wild-type, G551D, F508del, and R117H forms of human CFTR protein. Potentiators are pharmacological agents that increase the chloride ion transport properties of the channel in the presence of cyclic adenosine monophosphate (AMP)-dependent protein kinase A (PKA) activation.

DETAILED DESCRIPTION:
This study investigated the effects of ivacaftor in participants with cystic fibrosis (CF) >=12 years of age with a forced expiratory volume in 1 second (FEV1) >=40 percent (%) predicted. This study was conducted in 2 parts.

* Part A of this study was a randomized, double-blind, placebo-controlled, parallel-group evaluation of participants with CF who were aged 12 years or older and were homozygous for the F508del-CFTR mutation.
* Part B of this study was an open-label extension of Part A, enrolling participants who completed Part A and met pre-specified endpoint criteria, and explored the safety and efficacy of ivacaftor over long-term treatment in participants with CF aged 12 years or older who were homozygous for the F508del-CFTR mutation.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of cystic fibrosis (CF) and homozygous for F508del-CFTR mutation
* Forced expiratory volume in 1 second (FEV1) of at least 40% of predicted normal for age, gender, and height
* Willing to use at least 2 highly effective birth control methods during the study
* No clinically significant abnormalities that would have interfered with the study assessments, as judged by the investigator
* Able to understand and comply with protocol requirements, restrictions, and instructions and likely to complete the study as planned, as judged by the investigator

Exclusion Criteria:

* History of any illness or condition that might confound the results of the study or pose an additional risk in administering study drug to the subject
* Acute respiratory infection, pulmonary exacerbation, or changes in therapy for pulmonary disease within 4 weeks of Day 1 of the study
* History of alcohol, medication or illicit drug abuse within one year prior to Day 1
* Abnormal liver function >=3 x the upper limit of normal
* Abnormal renal function at Screening
* History of solid organ or hematological transplantation
* Pregnant or breast-feeding (for women)
* Ongoing participation in another therapeutic clinical study or prior participation in an investigational drug study within 30 days prior to screening
* Previous participation in a VX-809 study
* Used inhaled hypertonic saline treatment
* Concomitant use of any inhibitors or inducers of cytochrome P450 3A4 (CYP3A4)

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2009-09; Primary Completion 2010-07 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick A Flume, MD, Principal Investigator — Medical University of South Carolina
Locations (34):
- United States (34):
  - University of Alabama, Birmingham, Alabama
  - Providence Medical Center, Anchorage, Alaska
  - Kaiser Permanente Medical Care Program, Oakland, California
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - University of Miami Miller School of Medicine, Miami, Florida
  - Nemours Children's Clinic, Orlando, Florida
  - St. Luke's CF clinic, Boise, Idaho
  - University of Chicago, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Maine Medical Center, Portland, Maine
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Massachussetts Medical School, Worcester, Massachusetts
  - Helen DeVos Children's Hospital; Spectrum Health Hospitals, Grand Rapids, Michigan
  - The Children's Mercy Hospital, Kansas City, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Monmouth Medical Center, Long Branch, New Jersey
  - Morristown Memorial Hospital, Morristown, New Jersey
  - Albany Medical College, Albany, New York
  - Women and Children's Hospital of Buffalo, Buffalo, New York
  - New York Medical College, Hawthorne, New York
  - The CF Center, Beth Israel Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - Akron Children's Hospital, Akron, Ohio
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Toldedo Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Hershey Medical Center, Hershey, Pennsylvania
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Tennessee, Memphis, Tennessee
  - Cook Children's Medical Center, Fort Worth, Texas
  - Univeristy of Utah, Salt Lake City, Utah
  - Vermont Lung Center at the University of Vermont, Colchester, Vermont
  - Medical College of Virginia, Richmond, Virginia

REFERENCES:
- [Derived] Flume PA, Liou TG, Borowitz DS, Li H, Yen K, Ordonez CL, Geller DE; VX 08-770-104 Study Group. Ivacaftor in subjects with cystic fibrosis who are homozygous for the F508del-CFTR mutation. Chest. 2012 Sep;142(3):718-724. doi: 10.1378/chest.11-2672. PMID 22383668
- See also: Genetics Home Reference — http://ghr.nlm.nih.gov/handbook
- See also: Medline Plus — http://www.nlm.nih.gov/medlineplus/
- See also: U.S. FDA Resources — http://www.clinicaltrials.gov/ct2/info/fdalinks

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo - Part A: Placebo matched to ivacaftor tablet orally every 12 hours (q12h) for 16 weeks during Part A (double-blind treatment period).
- Ivacaftor - Part A: Ivacaftor 150 milligram (mg) tablet orally q12h for 16 weeks during Part A (double-blind treatment period).
- Placebo/Ivacaftor - Part B: Participants who received placebo during Part A, received ivacaftor 150 mg tablet orally q12h for 96 weeks during Part B (open-label extension period).
- Ivacaftor/Ivacaftor - Part B: Participants who received ivacaftor during Part A, received ivacaftor 150 mg tablet orally q12h for 96 weeks during Part B (open-label extension period).
Period: Part A (16-Week Double-Blind Treatment)
Arm/Group | Placebo - Part A | Ivacaftor - Part A | Placebo/Ivacaftor - Part B | Ivacaftor/Ivacaftor - Part B
Started | 28 (All subjects who received at least 1 dose of study drug (placebo)) | 112 (All subjects who received at least 1 dose of study drug (ivacaftor)) | 0 | 0
Completed | 26 (Only 5 participants continued in Part B.) | 104 (Only 33 participants continued in Part B.) | 0 | 0
Not Completed | 2 | 8 | 0 | 0
Not completed — Adverse Event | 2 | 3 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Noncompliance with Study Requirements | 0 | 2 | 0 | 0
Not completed — Required Prohibited Medication | 0 | 1 | 0 | 0
Not completed — Sponsor Decision | 0 | 1 | 0 | 0
Period: Part B (96-Week Open-Label Extension)
Arm/Group | Placebo - Part A | Ivacaftor - Part A | Placebo/Ivacaftor - Part B | Ivacaftor/Ivacaftor - Part B
Started | 0 | 0 | 5 | 33
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 5 | 33
Not completed — Adverse Event | 0 | 0 | 0 | 2
Not completed — Noncompliance with Study Requirements | 0 | 0 | 0 | 1
Not completed — Required Prohibited Medication | 0 | 0 | 0 | 1
Not completed — Study Termination by Sponsor | 0 | 0 | 4 | 25
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 2
Not completed — Other | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo - Part A | Ivacaftor - Part A | Total
Number analyzed (Participants) | 28 | 112 | 140
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.0 (8.35) | 22.8 (10.26) | 23.2 (9.91)
Age, Customized [Number; unit: participants]
  12 to 17 Years | 6 | 44 | 50
  18 to 24 Years | 10 | 32 | 42
  25 to 39 Years | 12 | 26 | 38
  40 to 45 Years | 0 | 5 | 5
  > 45 Years | 0 | 5 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 54 | 66
  Male | 16 | 58 | 74
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 27 | 110 | 137
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | 0 | 1 | 1
  White | 28 | 111 | 139
Percent Predicted Forced Expiratory Volume in 1 Second (ppFEV1), Continuous [Mean (Standard Deviation); unit: percent predicted of FEV1] — Percent predicted for age, gender, and height.
  percent predicted of FEV1 | 74.8 (24.06) | 79.7 (22.67) | 78.7 (22.95)
ppFEV1, Categorical [Number; unit: participants] — Percent predicted for age, gender, and height.
  participants
    < 70% | 15 | 38 | 53
    ≥ 70% to ≤ 90% | 5 | 35 | 40
    > 90% | 8 | 39 | 47
Weight [Mean (Standard Deviation); unit: kilograms] | 63.2 (14.96) | 58.2 (13.49) | 59.2 (13.89)
Body Mass Index [Mean (Standard Deviation); unit: kilogram per square meter] | 22.2 (4.48) | 21.2 (3.25) | 21.4 (3.54)
Sweat Chloride [Mean (Standard Deviation); unit: millimoles per liter] | 102.4 (7.91) | 101.4 (10.28) | 101.6 (9.83)

OUTCOME MEASURES:

1. Primary Outcome: Part A : Absolute Change From Part A Baseline in Percent Predicted Forced Expiratory Volume in 1 Second (ppFEV1) Through Week 16
Description: Spirometry (as measured by ppFEV1) is a standardized assessment to evaluate lung function that is the most widely used endpoint in cystic fibrosis studies. FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration. ppFEV1 (predicted for age, gender, and height) was calculated using the Knudson method.
Time Frame: Part A baseline through Week 16
Population: Part A Full Analysis Set (FAS) included all randomized participants who received at least 1 dose of study drug during Part A. Here, number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: percent predicted of FEV1
Groups:
- Placebo - Part A: Placebo matched to ivacaftor tablet orally q12h for 16 weeks during Part A (double-blind treatment period).
- Ivacaftor - Part A: Ivacaftor 150 mg tablet orally q12h for 16 weeks during Part A (double-blind treatment period).
Arm/Group | Placebo - Part A | Ivacaftor - Part A
Number analyzed (Participants) | 28 | 111
percent predicted of FEV1 | -0.2 (1.1) | 1.5 (0.5)
Statistical Analysis 1: Comparison: Placebo - Part A vs Ivacaftor - Part A; The primary analysis for the primary efficacy variable was based on a Mixed-Effects Model for Repeated Measures (MMRM). The model included absolute change from baseline in percent predicted forced expiratory volume in 1 second (FEV1) as the dependent variable, treatment (ivacaftor versus placebo) and visit as fixed effects, and participant as a random effect, with adjustment for age and continuous baseline value of percent predicted FEV1; Test type: Superiority or Other; p = 0.1509, Mixed Models Analysis; Mean Difference (Final Values) = 1.7, 95% CI 2-sided [-0.6 to 4.1], Standard Error of Mean 1.2

2. Secondary Outcome: Part A : Absolute Change From Part A Baseline in Cystic Fibrosis Questionnaire-Revised (CFQ-R) Respiratory Domain Score Through Week 16
Description: The CFQ-R is a validated patient-reported outcome measuring health-related quality of life for participants with cystic fibrosis. Respiratory domain assessed respiratory symptoms (for example, coughing, congestion, wheezing), score range: 0-100; Higher scores indicating fewer symptoms and better health-related quality of life.
Time Frame: Part A baseline through Week 16
Population: Part A FAS. Here, number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo - Part A | Ivacaftor - Part A
Number analyzed (Participants) | 28 | 111
units on a scale | -1.4 (1.9) | -0.1 (1.0)
Statistical Analysis 1: Comparison: Placebo - Part A vs Ivacaftor - Part A; Analysis for the respiratory domain score endpoint was similar to that of the primary analysis of the primary efficacy endpoint. Estimates were from Mixed-Effects Model for Repeated Measures (MMRM) with the dependent variable being absolute change from baseline, fixed effects for categorical visit and treatment group, and adjustment for for age and baseline value for CFQ-R score, using unstructured covariance matrix; Test type: Superiority or Other; p = 0.5408, Mixed Models Analysis; Mean Difference (Final Values) = 1.3, 95% CI 2-sided [-2.9 to 5.6], Standard Error of Mean 2.1

3. Secondary Outcome: Part A : Absolute Change From Part A Baseline in Sweat Chloride Concentration Through Week 16
Description: The sweat chloride (quantitative pilocarpine iontophoresis) test is a standard diagnostic tool for cystic fibrosis (CF), serving as an indicator of cystic fibrosis transmembrane conductance regulator (CFTR) activity.
Time Frame: Part A baseline through Week 16
Population: Part A FAS. Here, number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: millimole per liter (mmol/L)
Arm/Group | Placebo - Part A | Ivacaftor - Part A
Number analyzed (Participants) | 28 | 111
millimole per liter (mmol/L) | 0.1 (1.2) | -2.7 (0.6)
Statistical Analysis 1: Comparison: Placebo - Part A vs Ivacaftor - Part A; Analysis for this variable was similar to that of the primary analysis of the primary efficacy endpoint. Estimates were from Mixed-Effects Model for Repeated Measures (MMRM) with dependent variable being absolute change from baseline, fixed effects for categorical visit and treatment group, and adjustment for continuous age and baseline value for age, sweat chloride, using unstructured covariance matrix; Test type: Superiority or Other; p = 0.0384, Mixed Models Analysis; Mean Difference (Final Values) = -2.9, 95% CI 2-sided [-5.6 to -0.2], Standard Error of Mean 1.4

4. Secondary Outcome: Part A : Rate of Change From Baseline in Weight Through Week 16
Description: As malnutrition is common in participants with cystic fibrosis (CF) because of increased energy expenditures due to lung disease and fat malabsorption, body weight is an important clinical measure of nutritional status.
Time Frame: Part A baseline through Week 16
Population: Part A FAS. Here, number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: kilograms per 112 days
Arm/Group | Placebo - Part A | Ivacaftor - Part A
Number analyzed (Participants) | 28 | 112
kilograms per 112 days | 0.9 (0.4) | 0.8 (0.2)
Statistical Analysis 1: Comparison: Placebo - Part A vs Ivacaftor - Part A; The analysis used the linear mixed model with treatment as fixed effects, visit (days on study) and treatment by visit interaction as random effects, with adjustment for age group (< 18 years and ≥ 18 years) and percent predicted forced expiratory volume (FEV1) severity (< 70%, ≥ 70% to ≤ 90%, > 90%) at screening, with random intercept and random slope. Rate of change in the study period is the slope of weight versus time (days) multiplied by the number of days in the study period (112 days); Test type: Superiority or Other; p = 0.7265, Mixed Models Analysis; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-1.1 to 0.7], Standard Error of Mean 0.5

5. Secondary Outcome: Part B : Absolute Change From Part A and Part B Baseline in ppFEV1 Through Week 64
Description: ppFEV1 is defined in Outcome Measure 1.
Time Frame: Change from Part A baseline: Part A Baseline, Week 64; Change from Part B baseline: Part B Baseline (Week 16), Week 64
Population: Part B FAS included all participants who received at least 1 dose of study drug during Part B. Here, number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: percent predicted of FEV1
Arm/Group | Placebo/Ivacaftor - Part B | Ivacaftor/Ivacaftor - Part B
Number analyzed (Participants) | 4 | 27
percent predicted of FEV1
  Change From Part A Baseline at Week 64 | 8.9398 (9.70300) | 2.7233 (10.52046)
  Change From Part B Baseline at Week 64 | 3.5593 (7.95875) | -5.0565 (11.44783)

6. Secondary Outcome: Part B : Rate of Change From Part A Baseline in ppFEV1 Through Week 64
Description: ppFEV1 is defined in Outcome Measure 1.
Time Frame: Part A baseline through Week 64
Population: Part B FAS.
Measure: Least Squares Mean (Standard Error); unit: percent predicted of FEV1 per 448 days
Arm/Group | Placebo/Ivacaftor - Part B | Ivacaftor/Ivacaftor - Part B
Number analyzed (Participants) | 5 | 33
percent predicted of FEV1 per 448 days | 5.7445 (3.6810) | -1.0738 (1.5025)

7. Secondary Outcome: Part B : Rate of Change From Part B Baseline in ppFEV1 Through Week 64
Description: ppFEV1 is defined in Outcome Measure 1.
Time Frame: Part B baseline through Week 64
Population: Part B FAS.
Measure: Least Squares Mean (Standard Error); unit: percent predicted of FEV1 per 336 days
Arm/Group | Placebo/Ivacaftor - Part B | Ivacaftor/Ivacaftor - Part B
Number analyzed (Participants) | 5 | 33
percent predicted of FEV1 per 336 days | 5.3409 (4.5790) | -5.2994 (1.8871)

8. Secondary Outcome: Part B : Absolute Change From Part A and Part B Baseline in CFQ-R Respiratory Domain Score Through Week 64
Description: as for outcome 2
Time Frame: Change from Part A baseline: Part A Baseline, Week 64; Change from Part B baseline: Part B Baseline (Week 16), Week 64
Population: Part B FAS. Here, number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo/Ivacaftor - Part B | Ivacaftor/Ivacaftor - Part B
Number analyzed (Participants) | 4 | 26
units on a scale
  Change From Part A Baseline at Week 64 | 2.10 (11.443) | 1.50 (15.778)
  Change From Part B Baseline at Week 64 | 2.08 (17.763) | 2.62 (15.899)

9. Secondary Outcome: Part B : Absolute Change From Part A and Part B Baseline in Sweat Chloride Concentration Through Week 64
Description: as for outcome 3
Time Frame: Change from Part A baseline: Part A Baseline, Week 64; Change from Part B baseline: Part B Baseline (Week 16), Week 64
Population: Part B FAS. Here, number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo/Ivacaftor - Part B | Ivacaftor/Ivacaftor - Part B
Number analyzed (Participants) | 4 | 26
mmol/L
  Change From Part A Baseline at Week 64 | -7.13 (15.612) | -3.65 (11.963)
  Change From Part B Baseline at Week 64 | -3.88 (7.685) | -2.44 (11.037)

10. Secondary Outcome: Part B : Absolute Change From Part A and Part B Baseline in Weight Through Week 64
Description: As malnutrition is common in patients with cystic fibrosis (CF) because of increased energy expenditures due to lung disease and fat malabsorption, body weight is an important clinical measure of nutritional status.
Time Frame: Change from Part A baseline: Part A Baseline, Week 64; Change from Part B baseline: Part B Baseline (Week 16), Week 64
Population: Part B FAS. Here, number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: kilograms (kg)
Arm/Group | Placebo/Ivacaftor - Part B | Ivacaftor/Ivacaftor - Part B
Number analyzed (Participants) | 4 | 27
kilograms (kg)
  Change From Part A Baseline at Week 64 | 3.00 (3.550) | 2.35 (5.600)
  Change From Part B Baseline at Week 64 | 1.28 (2.243) | 1.45 (3.840)

11. Secondary Outcome: Part B : Number of Participants With Pulmonary Exacerbations
Description: Pulmonary exacerbation was defined as new, or changed, antibiotic therapy (intravenous, inhaled, or oral) for any 4 or more of the following signs/symptoms: change in sputum; new or increased hemoptysis; increased cough; increased dyspnea; malaise, fatigue, or lethargy; temperature above 38 degrees Celsius; anorexia or weight loss; sinus pain or tenderness; change in sinus discharge; change in physical examination of the chest; decrease in pulmonary function by 10 percent (%); and radiographic changes indicative of pulmonary infection.
Time Frame: Part B baseline through Week 64
Population: Part B FAS.
Measure: Number; unit: participants
Arm/Group | Placebo/Ivacaftor - Part B | Ivacaftor/Ivacaftor - Part B
Number analyzed (Participants) | 5 | 33
participants | 4 | 16

12. Secondary Outcome: Part B : Number of Pulmonary Exacerbation Events
Description: as for outcome 11
Time Frame: Part B baseline through Week 64
Population: Part B FAS.
Measure: Number; unit: events
Arm/Group | Placebo/Ivacaftor - Part B | Ivacaftor/Ivacaftor - Part B
Number analyzed (Participants) | 5 | 33
events | 6 | 26

13. Secondary Outcome: Part B : Number of Pulmonary Exacerbation Events Per Participant Per Year
Description: as for outcome 11
Time Frame: Part B baseline through Week 64
Population: Part B FAS.
Measure: Number; unit: events per participant per year
Arm/Group | Placebo/Ivacaftor - Part B | Ivacaftor/Ivacaftor - Part B
Number analyzed (Participants) | 5 | 33
events per participant per year | 1.10 | 0.82

ADVERSE EVENTS:
Time Frame: Adverse events (serious and non-serious) were collected from signing of informed consent through 2 years after last dose (in Part B) of study drug (median treatment duration: 112 days for Part A and 381 days for Part B)
Arm/Group | Placebo - Part A | Ivacaftor - Part A | Placebo/Ivacaftor - Part B | Ivacaftor/Ivacaftor - Part B
Serious Adverse Events (participants affected / at risk) | 6/28 | 15/112 | 2/5 | 14/33
Other Adverse Events (participants affected / at risk) | 25/28 | 98/112 | 5/5 | 30/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo - Part A (N=28) | Ivacaftor - Part A (N=112) | Placebo/Ivacaftor - Part B (N=5) | Ivacaftor/Ivacaftor - Part B (N=33)
Cystic fibrosis lung (Congenital, familial and genetic disorders) | 5 (6) | 10 (12) | 2 (4) | 13 (20) — CF exacerbations were coded as "cystic fibrosis lung."
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchopneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Central line infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Traumatic brain injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Venous thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo - Part A (N=28) | Ivacaftor - Part A (N=112) | Placebo/Ivacaftor - Part B (N=5) | Ivacaftor/Ivacaftor - Part B (N=33)
Cystic fibrosis lung (Congenital, familial and genetic disorders) | 7 (8) | 19 (24) | 3 (6) | 11 (17) — CF exacerbations were coded as "cystic fibrosis lung."
Abdominal pain upper (Gastrointestinal disorders) | 1 (4) | 7 (8) | 0 (0) | 2 (3)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 6 (7) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 10 (11) | 0 (0) | 3 (3)
Chills (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 3 (3) | 8 (8) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 9 (10) | 0 (0) | 2 (3)
Acute sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Clostridium Difficile colitis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 4 (5) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Orchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pneumonia staphylococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory monilliasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 5 (5) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 8 (9) | 1 (1) | 4 (5)
Stenotrophomonas infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tinea infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 11 (13) | 1 (1) | 1 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
Alanine aminotransferase increased (Investigations) | 2 (3) | 1 (1) | 0 (0) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 2 (3) | 1 (1) | 0 (0) | 1 (1)
C-reactive protein increased (Investigations) | 1 (1) | 6 (6) | 0 (0) | 0 (0)
Pulmonary function test decreased (Investigations) | 2 (2) | 3 (4) | 0 (0) | 1 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 0 (0) | 3 (3)
Dizziness (Nervous system disorders) | 2 (2) | 2 (3) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (3) | 11 (17) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 34 (43) | 0 (0) | 15 (17)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5) | 1 (1) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (10) | 2 (3) | 2 (2)
Increased viscosity of bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 13 (14) | 0 (0) | 2 (2)
Nasal mucosal disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Nasal oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 10 (12) | 0 (0) | 1 (1)
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngeal disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 9 (9) | 0 (0) | 4 (5)
Rales (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (4) | 0 (0) | 2 (2)
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (4) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (5) | 0 (0) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 6 (9) | 0 (0) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 9 (9) | 0 (0) | 1 (1)
Bacterial disease carrier (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Body tinea (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Helicobacter gastritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infectious mononucleosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaginitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 1 (1) | 5 (5) | 0 (0) | 1 (1)
Bacteria sputum identified (Investigations) | 1 (1) | 3 (4) | 0 (0) | 1 (1)
Prothrombin time prolonged (Investigations) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Gamma-glutamyl transferase increased (Investigations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Glucose urine present (Investigations) | 0 (0) | 3 (4) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Blood immunoglobulin G increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Breath sounds abnormal (Investigations) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Forced expiratory volume decreased (Investigations) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Vitamin D decreased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Acivated partial thromboplastin time prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Antibiotic level above therapeutic (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bacterial culture positive (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood glucose decreased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Bone density decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Liver function test abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sputum culture positive (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Oxygen saturation decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sputum abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 4 (5) | 3 (3) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aphthous stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (2)
Dental Caries (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Distal Ileal Obstruction Syndrome (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Dry Mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Frequent Bowel Movements (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Gastrointestinal Hypomotility (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hiatus Hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pancreatic Duct Dilatation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peptic Ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Regurgitation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth Impacted (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Distal Intestinal Obstruction Syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sensitivity Of Teeth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catheter Site Pain (General disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Application Site Pruritus (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Application Site Rash (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Feeling Abnormal (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Generalised Oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza Like Illness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thirst (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vessel Puncture Site Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Catheter Related Complication (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion Site Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema Peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cystic Fibrosis Related Diabetes (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Rash Papular (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Rash Vesicular (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Night Sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Photodermatosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Photosensitivity Reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rash Macular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 2 (3)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Red Man Syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Sinus Headache (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Burning Sensation (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (5) | 0 (0) | 4 (4)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 2 (2) | 0 (0) | 2 (3)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 2 (3)
Joint Swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Clubbing (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Synovial Cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 2 (3) | 0 (0) | 1 (1)
Skin Laceration (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Foreign Body Trauma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint Sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle Strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Procedural Pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural Site Reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thermal Burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Traumatic Brain Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Animal Bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Arthropod Sting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Head Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Lacrimation Increased (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis Allergic (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye Pruritus (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eyelid Oedema (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Visual Impairment (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erythema Of Eyelid (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 0 (0) | 2 (2)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vitamin D Deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Glucose Tolerance Impaired (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypovitaminosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Abnormal Dreams (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
Hallucination (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adjustment Disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Calculus Bladder (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chromaturia (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal Cyst (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal Failure Acute (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast Tenderness (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prostatic Cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Testicular Pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Testicular Swelling (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Middle Ear Effusion (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatosplenomegaly (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Allergy to Animal (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Seasonal Allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Supraventricular Extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Focal Nodular Hyperplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
wisdom teeth removal (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
In Part B, the treatment duration was 96 weeks; however, due to early study termination all analysis were performed up to Week 64, as planned.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days